CLINICAL TRIAL: NCT06774729
Title: Development of a Radiomics Model With 3T Multiparametric MR to Predict the Occurence of a Perilesional Infiltration of Muscoskeletal Tumor During the Pre- Surgery Planning
Brief Title: Development of a Radiomics Model With MR to Predict the Occurence of a Infiltration of Muscoskeletal Tumor
Status: Recruiting | Type: Observational
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Responsible Party: Sponsor
Other Study IDs: MIT3
Record Dates: First submitted 2025-01-09; First posted 2025-01-14 (Actual); Last update posted 2025-01-14 (Actual); Status verified 2024-10

CONDITIONS: Soft Tissue Sarcoma (STS); Bone Cancer Tumor
MeSH Terms: conditions — Sarcoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this observational study is to evaluate the feasibility and clinical utility of radiomics to diagnose peri-lesion tumour infiltration of tumours in participants with a suspect of Bone Cancer Tumor or Soft Tissue Sarcoma (STS).

The main questions it aims to answer are:

* is radiomics able to identify the ratio of participants truly diagnosed as positive to all those who had positive test results?
* is radiomics able to identify the likelihood that a participant who has a negative test result indeed does not have the disease?

Participants eligible for this study will get a MRI as part of their regular medical care. The only difference is that their data will be recorded and anonymously analyzed.

ELIGIBILITY:
Inclusion Criteria:

* Age over 18
* suspect of soft tissue sarcoma with a indication for surgical treatment
* suspect of bone cancer tumor with a indication for surgical treatment
* To give informed consent

Exclusion Criteria:

* simultaneous cancer or history of cancer in the last 5 years
* acute or chronic serious conditions that could
* contraindication to conduct a Contrast-enhanced magnetic resonance imaging (MRI) such as:

  * renal failure without dialysis
  * history of allergy to a paramagnetic contrast agent
  * claustrophobia
  * symptomatic epilepsy or history of epilepsy
  * cardiac pacemaker
  * infusion pump, prosthesis or any implant not compatible with MRI
  * pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population consists in participants with a suspect of soft tissue sarcoma or bone cancer that are followed at Radiology Department of IRCCS Azienda Ospedaliero-Universitaria hospital in the city of Bologna.
Sampling Method: Non-Probability Sample
Enrollment: 122 (Estimated)
Dates: Start 2025-03 (Estimated); Primary Completion 2028-09 (Estimated); Study Completion 2028-10 (Estimated)

PRIMARY OUTCOMES:
Positive Predictive Value (PPV) | From enrollment to the end of treatment at 2 years
  It is the ratio of patients truly diagnosed as positive to all those who had positive test results (including healthy subjects who were incorrectly diagnosed as patient).
Negative Predictive Value (NPV) | From enrollment to the end of treatment at 2 years
  It is the ratio of subjects truly diagnosed as negative to all those who had negative test results (including patients who were incorrectly diagnosed as healthy).

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS Azienda Ospedaliero-Universitaria di Bologna, Bologna, Italy